CLINICAL TRIAL: NCT06823219
Title: Evaluation of a Long-term Endurance Training Program in Patients With Sickle Cell Disease: Benefits on Clinical Profile, Physical Fitness and Quality of Life of Patients
Brief Title: Long-term Endurance Training in Sickle Cell Disease Patients: Impact on Clinical Profile, Physical Fitness, and Quality of Life.
Acronym: EXDRE2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP230822
Record Dates: First submitted 2024-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; , endurance training
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, controlled trial, multicentric, open label
Masking Description: Randomization will be in a 1:2 ratio between the untrained and trained arms, respectively. Randomization will be stratified on treatment by hydroxyurea, gender and age.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trained arm (Experimental): Groupe 2: 52 weeks of out-of-hospital physical activity (The patients of the trained arm with a V̇O2 at SL2 >75% of the predicted V̇O2 at SL2) Groupe 3: 8 weeks of in hospital endurance training 3/weeks and 44 weeks of out- of-hospital physical activity (Patients identified as presenting severity criteria )
  Interventions: Other: endurance training program
- untrained arm (No Intervention): Groupe 1: 52 weeks of unchanged rhythm

INTERVENTIONS:
Other: endurance training program — Groupe 2: 52 weeks of out-of-hospital physical activity Groupe 3: 8 weeks of in hospital endurance training 3/weeks and 44 weeks of out- of-hospital physical activity
  Arms: trained arm

SUMMARY:
Sickle cell disease (SCD), the most common genetic disease worldwide and in France, is an inherited haemoglobinopathy characterised by chronic haemolytic anaemia, vaso-occlusive crisis (VOC), acute pain, and multi-organ damage. Due to anaemia and multiple pulmonary, cardiac, endothelial, muscle, and metabolic dysfunctions, fatigue and poor physical capacity are common in SCD patients and constitute the primary reason for a sedentary lifestyle.

However, recent findings demonstrated in the first randomised, controlled, and prospective study implementing endurance training in SCD that, when adequately calibrated, regular moderate-intensity endurance training is not only safe but also beneficial for patients (primary outcome: improvement of physical ability).

This pivotal randomised, controlled, prospective study is designed to prove, on a large multicentre cohort, adult and paediatric, including patients with complications and over a longer period (one year).

The objective of the study is to demonstrate the efficacy of participating in a program of regular physical activity to reduce the rate of vaso-occlusive crises requiring hospitalisation and to improve physical ability in patients with SCD.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is an inherited haemoglobinopathy characterised by chronic haemolytic anaemia, vaso-occlusive crisis (VOC), acute pain, and multi-organ damage, making it the most common genetic disease in France. The mutation involves the substitution of glutamic acid by valine at position β6, leading to the synthesis of abnormal haemoglobin (HbS). The properties of HbS differ significantly from those of normal haemoglobin (HbA). Under deoxygenated conditions, HbS tends to polymerize, inducing deformation of the red blood cell (RBC), causing it to take on a sickle shape.

This leads to a very low haemoglobin concentration and haematocrit (typically 6-8 g/dL and 25%-30%, respectively). Anaemia, coupled with arterial desaturation, results in tissue hypoxia. Furthermore, RBCs containing HbS (RBC-HbS) are less deformable and exhibit abnormal adherence properties. The reduced deformability of HbS-containing RBCs, along with the stiffening of sickle-shaped RBCs, impedes their passage through small vessels, potentially causing blockages in capillaries and obstructing microcirculation, leading to the particularly painful vaso-occlusive crisis (VOC).

In patients with SCD, physical exercise has been shown to be physiologically stressful, resulting in severe exercise intolerance.

Exercise limitations in SCD are related to anaemia, as walking for 5 minutes at 5 km/h leads to large elevations in heart rate (~175 beats/min) and blood lactate concentration (6.6 ± 0.4 mmol/L) in patients. This indicates that exercise, which is relatively easy for sedentary healthy adults, is already too difficult for patients with SCD. Additionally, the first lactate threshold is around 30-35 W for women and 44-50 W for men. These extremely low values reflect the significantly reduced physical ability of patients with SCD, suggesting that even common daily tasks are challenging for them.

The National Sports Health Strategy (SNSS) promotes physical activity for chronic conditions, including SCD.

This project aligns with the second axis of the SNSS, which focuses on the development and use of adapted physical activity as a therapeutic treatment for SCD patients.

Endurance training for trained groups involves a submaximal incremental cycling test. The total test duration is expected to range from 9 to 15 minutes. During the last 5 seconds of each step, a blood sample (7 µL) will be taken from the earlobe and immediately analysed (in less than 20 seconds using Lactate Scout+, EKF Diagnostics) to determine the blood lactate concentration ([lactate]b). Exercise should cease when a [lactate]b of 4 mmol/L is reached. This protocol will allow for the determination of exercise powers and heart rates at the first lactate threshold, at 2.5 mmol/L, and at 4 mmol/L. These values will help set the heart rates used during training/physical activity and assess the physical fitness of patients.

The study will occur in four main stages:

i) A screening visit ii) An initial evaluation of the patients (W0, Initial Evaluations), which includes two visits: an inclusion visit (V0) and a physical evaluation visit (V1) iii) A 52-week period (W1-W52) where the control group maintains their usual inactive lifestyle, while the trained groups engage in training and/or physical activity following a therapeutic education session (V2apa) iv) The period will be interspersed with evaluations at M6/W25 and followed by evaluations at M12/W52. These evaluations will include two visits (V3 and V4 at M6, and V5 and V6 at M12), similar to V0 and V1.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 15 years and 3 months
* Male or female
* Patients with sickle cell disease (HbSS or HbS-βthal0)
* Affiliated to a social security system
* Having freely given their written consent after having been informed of the purpose, the procedure and the potential risks involved
* Patients in stabilised condition at the start of the experiment: at least 1 month after an acute chronic event or at least 3 months after a blood transfusion.
* Patients hospitalised for vaso-occlusive crisis at least once in the last 3 years

Exclusion Criteria:

* Patient whose adherence to the protocol is unlikely according to the investigator
* Patients who already partake in regular physical activity (more than 1 hour of moderate-intensity physical activity per week)
* Patients with a chronic inflammatory and/or infectious pathology
* Patients with an intercurrent condition unresolved for less than a month
* Patients hospitalised for cardiac decompensation during the last 12 months
* Patients on anticoagulant treatment or with a pacemaker/defibrillator
* Pregnant patients / breastfeeding woman
* Patients deprived of liberty by judicial or administrative decision or patient under guardianship
* Patients unable to understand the objectives and conditions of the study and unable to give cons

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of vaso-occlusive crises (VOCs) with hospitalisation | 12 months
  determine the hospitalization rate for vaso-occlusive crisis
Exercise capacity and muscle metabolism and characteristics | 12 months
  the change from baseline in the workload at first lactate threshold. A blood sample (7 µL) will be taken from the earlobe and immediately analysed (in less than 20 seconds, Lactate Scout+, EKF Diagnostics) to determine the blood lactate concentration ([lactate]b). Exercise should be stopped when a [lactate]b of 4 mmol/L is reached

SECONDARY OUTCOMES:
Duration of hospitalisation | 12 months
Median time from the initiation of "treatment" (training or habitual (inactive) lifestyle) to the first and second hospitalised VOC | 12 months
Number of acute chest syndromes (ACS) | 12 months
Days of school and job absenteeism | 12 months
Analgesic intake | 12 months
6-minute walk test (6MWT) - performed | 12 months
  The 6MWT will assess the endurance and functional capacities of patients. Distance at 6MWT completion will be measured, as well as the time spent under 90% of oxygen saturation during the test. The patients' Rating of Perceived Exertion (RPE) using the 0-10 Borg's scale will be recorded
Echocardiographic Parameters | 12 months
  Left ventricular ejection fraction (LVEF) (%)
Echocardiographic Parameters | 12 months
  Ventricular wall motion (qualitative assessment or mm)
Echocardiographic Parameters | 12 months
  Chamber Dimensions (mm or mL)
Exercise Physiology Parameters | 12 months
  Heart rate (HR) (beats per minute - bpm)

CONTACTS AND LOCATIONS:
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No